CLINICAL TRIAL: NCT05489328
Title: A PHASE 1, RANDOMIZED, OPEN-LABEL TRIAL TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF PNEUMOCOCCAL CONJUGATE FORMULATIONS IN HEALTHY ADULTS 18 THROUGH 49 YEARS OF AGE
Brief Title: Safety and Immunogenicity of Pneumococcal Conjugate Formulations in Healthy Adults 18 Through 49 Years of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C4801001
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Candidate-1 (Experimental): Participants to receive a single injection of Candidate-1.
  Interventions: Other: Candidate-1
- Candidate-2 (Experimental): Participants to receive a single injection of Candidate-2.
  Interventions: Other: Candidate-2
- Candidate-3 (Experimental): Participants to receive a single injection of Candidate-3.
  Interventions: Other: Candidate-3
- Candidate-4 (Experimental): Participants to receive a single injection of Candidate-4.
  Interventions: Other: Candidate-4
- Candidate-5 (Experimental): Participants to receive a single injection of Candidate-5.
  Interventions: Other: Candidate-5
- Candidate-6 (Experimental): Participants to receive a single injection of Candidate-6.
  Interventions: Other: Candidate-6
- Candidate Control (Active Comparator): Participants to receive a single injection of Candidate Control.
  Interventions: Other: Candidate Control
- 13-valent pneumococcal conjugate vaccine (13vPnC) (Other): Participants to receive a single injection of 13vPnC.
  Interventions: Biological: 13vPnC
- 15-valent pneumococcal conjugate vaccine (PCV15) (Other): Participants to receive a single injection of PCV15.
  Interventions: Biological: PCV15

INTERVENTIONS:
Other: Candidate-1 — Biological
  Arms: Candidate-1
Other: Candidate-2 — Biological
  Arms: Candidate-2
Other: Candidate-3 — Biological
  Arms: Candidate-3
Other: Candidate-4 — Biological
  Arms: Candidate-4
Other: Candidate-5 — Biological
  Arms: Candidate-5
Other: Candidate-6 — Biological
  Arms: Candidate-6
Other: Candidate Control — Biological
  Arms: Candidate Control
Biological: 13vPnC — 13-valent pneumococcal conjugate vaccine
  Arms: 13-valent pneumococcal conjugate vaccine (13vPnC)
Biological: PCV15 — 15-valent pneumococcal conjugate vaccine
  Arms: 15-valent pneumococcal conjugate vaccine (PCV15)

SUMMARY:
The purpose of the study is to describe the safety and immunogenicity of Pneumococcal Conjugate Formulations in healthy adults 18 through 49 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥18 and ≤49 years of age at the time of consent
* Adults determined by clinical assessment to be eligible for the study, including adults with preexisting stable disease within 12 weeks before receipt of study intervention
* Participants willing to use acceptable contraception for at least 28 days after study intervention; female participants not of childbearing potential; male participants unable to father children

Exclusion Criteria:

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction to any component in pneumococcal conjugate vaccines and any other diphtheria toxoid-containing vaccine
* Serious chronic disorder that in the investigator's opinion would make the participant inappropriate for entry into the study
* Medical or psychiatric condition (recent or active suicidal ideation/behavior or laboratory abnormality) that may increase risk of study participation or make participant inappropriate for the study
* Known or suspected immunodeficiency or other conditions associated with immunosuppression
* Previous vaccination with any licensed or investigational pneumococcal vaccine, or planned receipt of any licensed or investigational pneumococcal vaccine through study participation
* Receipt of any inactivated or otherwise nonlive vaccine within 14 days or any live vaccine within 28 days before administration of study intervention

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 394 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- United States (18):
  - Orange County Research Center, Tustin, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Clinical Research Consulting, Milford, Connecticut
  - Proactive Clinical Research,LLC, Fort Lauderdale, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Qps-Mra, Llc, South Miami, Florida
  - Centennial Medical Group, Elkridge, Maryland
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - Prism Research LLC dba Nucleus Network, Saint Paul, Minnesota
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Accellacare - Wilmington, Wilmington, North Carolina
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
  - DM Clinical Research, Tomball, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - Alliance for Multispecialty Research, LLC, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4801001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 17 sites in the United States.
Pre-assignment Details: A total of 394 participants were enrolled and randomized in the study of which 3 participants were not vaccinated and, 391 were administered study intervention. One participant randomized to Candidate-Control received Candidate-4.
Groups:
- Candidate-1: Participants were administered a single intramuscular injection of candidate-1 on Day 1. Participants were followed up for 1 month (28-42 days) after administration of study intervention.
- Candidate-2: Participants were administered a single intramuscular injection of candidate-2 on Day 1. Participants were followed up for 1 month (28-42 days) after administration of study intervention.
- Candidate-3: Participants were administered a single intramuscular injection of candidate-3 on Day 1. Participants were followed up for 1 month (28-42 days) after administration of study intervention.
- Candidate-4: Participants were administered a single intramuscular injection of candidate-4 on Day 1. Participants were followed up for 1 month (28-42 days) after administration of study intervention.
- Candidate-5: Participants were administered a single intramuscular injection of candidate-5 on Day 1. Participants were followed up for 1 month (28-42 days) after administration of study intervention.
- Candidate-6: Participants were administered a single intramuscular injection of candidate-6 on Day 1. Participants were followed up for 1 month (28-42 days) after administration of study intervention.
- Candidate - Control: Participants were administered a single intramuscular injection of control on Day 1. Participants were followed up for 1 month (28-42 days) after administration of study intervention.
- PCV15: Participants were administered a single intramuscular injection of pneumococcal 15-valent conjugate (PCV15) vaccine (control) on Day 1. Participants were followed up for 1 month (28-42 days) after administration of study intervention.
- 13vPnC: Participants were administered a single intramuscular injection of Prevnar 13 vaccine (control) on Day 1. Participants were followed up for 1 month (28-42 days) after administration of study intervention.
Period: Overall Study
Arm/Group | Candidate-1 | Candidate-2 | Candidate-3 | Candidate-4 | Candidate-5 | Candidate-6 | Candidate - Control | PCV15 | 13vPnC
Started (Participants who were randomized) | 41 | 42 | 39 | 43 | 45 | 46 | 47 | 44 | 47
Vaccinated (Participants who were administered the study intervention) | 41 | 42 | 39 | 43 | 45 | 46 | 46 (One participant received Candidate-4.) | 43 | 46
Completed | 41 | 42 | 38 | 43 | 43 | 46 | 46 | 41 | 46
Not Completed | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 3 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety population which included all participants who received the study intervention. Participants were summarized according to the study intervention they received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Candidate-1 | Candidate-2 | Candidate-3 | Candidate-4 | Candidate-5 | Candidate-6 | Candidate - Control | PCV15 | 13vPnC | Total
Number analyzed (Participants) | 41 | 42 | 39 | 44 | 45 | 46 | 45 | 43 | 46 | 391
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.9 (9.15) | 35.2 (9.11) | 35.3 (9.44) | 33.2 (9.39) | 33.3 (9.29) | 35.2 (8.35) | 34.1 (7.68) | 35.6 (8.86) | 35.7 (7.38) | 34.8 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 26 | 27 | 24 | 26 | 25 | 27 | 19 | 23 | 227
  Male | 11 | 16 | 12 | 20 | 19 | 21 | 18 | 24 | 23 | 164
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 15 | 12 | 12 | 12 | 20 | 14 | 14 | 16 | 128
  Not Hispanic or Latino | 27 | 27 | 27 | 32 | 33 | 26 | 31 | 29 | 30 | 262
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  Asian | 1 | 2 | 3 | 3 | 3 | 1 | 4 | 1 | 4 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Black or African American | 14 | 4 | 8 | 8 | 5 | 6 | 9 | 7 | 8 | 69
  White | 25 | 35 | 26 | 32 | 36 | 37 | 30 | 33 | 32 | 286
  More than one race | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Administration of Study Intervention
Description: Local reactions included redness, swelling and pain at the injection site collected in an electronic diary (e-diary) or case report form(CRF). Redness and swelling were measured and recorded in measuring device units. One measuring device unit=0.5 centimeter (cm). Redness and swelling reported in e-diary were graded as mild: greater than (>) 2.0 cm to 5.0 cm, moderate: >5.0 cm to 10.0 cm and severe > 10 cm. Pain at injection site was graded as mild: did not interfere with activity; moderate: interfered with activity; and severe: prevented daily activity. Severity definition from CRF: mild (does not interfere)/moderate (interferes to some extent)/severe(interferes significantly) with the participant's usual function. Exact 2-sided 95% confidence interval (CI) was based on the Clopper and Pearson method.
Time Frame: Within 7 days after study intervention
Population: Safety population included all participants who received the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Candidate-1 | Candidate-2 | Candidate-3 | Candidate-4 | Candidate-5 | Candidate-6 | Candidate - Control | PCV15 | 13vPnC
Number analyzed (Participants) | 41 | 42 | 39 | 44 | 45 | 46 | 45 | 43 | 46
Percentage of participants
  Redness: Mild | 0.0 [0.0 to 8.6] | 0.0 [0.0 to 8.4] | 0.0 [0.0 to 9.0] | 2.3 [0.1 to 12.0] | 2.2 [0.1 to 11.8] | 4.3 [0.5 to 14.8] | 0.0 [0.0 to 7.9] | 4.7 [0.6 to 15.8] | 0.0 [0.0 to 7.7]
  Redness: Moderate | 0.0 [0.0 to 8.6] | 2.4 [0.1 to 12.6] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.0] | 2.2 [0.1 to 11.8] | 2.2 [0.1 to 11.5] | 0.0 [0.0 to 7.9] | 4.7 [0.6 to 15.8] | 2.2 [0.1 to 11.5]
  Redness: Severe | 0.0 [0.0 to 8.6] | 0.0 [0.0 to 8.4] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 8.2] | 0.0 [0.0 to 7.7]
  Swelling: Mild | 0.0 [0.0 to 8.6] | 0.0 [0.0 to 8.4] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.0] | 2.2 [0.1 to 11.8] | 6.5 [1.4 to 17.9] | 0.0 [0.0 to 7.9] | 4.7 [0.6 to 15.8] | 8.7 [2.4 to 20.8]
  Swelling: Moderate | 0.0 [0.0 to 8.6] | 2.4 [0.1 to 12.6] | 0.0 [0.0 to 9.0] | 2.3 [0.1 to 12.0] | 2.2 [0.1 to 11.8] | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 7.9] | 4.7 [0.6 to 15.8] | 0.0 [0.0 to 7.7]
  Swelling: Severe | 0.0 [0.0 to 8.6] | 0.0 [0.0 to 8.4] | 2.6 [0.1 to 13.5] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 7.9] | 2.2 [0.1 to 11.5] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 8.2] | 0.0 [0.0 to 7.7]
  Pain At Injection Site: Mild | 12.2 [4.1 to 26.2] | 26.2 [13.9 to 42.0] | 20.5 [9.3 to 36.5] | 25.0 [13.2 to 40.3] | 37.8 [23.8 to 53.5] | 23.9 [12.6 to 38.8] | 11.1 [3.7 to 24.1] | 37.2 [23.0 to 53.3] | 54.3 [39.0 to 69.1]
  Pain At Injection Site: Moderate | 0.0 [0.0 to 8.6] | 4.8 [0.6 to 16.2] | 0.0 [0.0 to 9.0] | 2.3 [0.1 to 12.0] | 6.7 [1.4 to 18.3] | 17.4 [7.8 to 31.4] | 2.2 [0.1 to 11.8] | 30.2 [17.2 to 46.1] | 6.5 [1.4 to 17.9]
  Pain At Injection Site: Severe | 0.0 [0.0 to 8.6] | 0.0 [0.0 to 8.4] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 8.2] | 2.2 [0.1 to 11.5]

2. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Administration of Study Intervention
Description: Systemic events included fever, fatigue, headache, muscle pain and joint pain and were collected in an e-diary or CRF. Fever was defined as temperature greater than or equal to (>=) 38.0 degrees Celsius (C) and categorized as >=38.0 to 38.4 degrees C, >38.4 to 38.9 degrees C, >38.9 to 40.0 degrees C and >40.0 degrees C. Fatigue, headache, muscle pain and joint pain were graded as mild: did not interfere with activity; moderate: some interference with activity and severe: prevented daily routine activities. Severity definition from the CRF: mild (does not interfere)/moderate(interferes to some extent)/severe(interferes significantly) with the participant's usual function. Exact 2-sided 95% CI was based on the Clopper and Pearson method.
Time Frame: Within 7 days after study intervention
Population: Safety population included all participants who received the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Candidate-1 | Candidate-2 | Candidate-3 | Candidate-4 | Candidate-5 | Candidate-6 | Candidate - Control | PCV15 | 13vPnC
Number analyzed (Participants) | 41 | 42 | 39 | 44 | 45 | 46 | 45 | 43 | 46
Percentage of participants
  Fever: >/=38.0 degrees C to 38.4 degrees C | 0.0 [0.0 to 8.6] | 0.0 [0.0 to 8.4] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.0] | 2.2 [0.1 to 11.8] | 4.3 [0.5 to 14.8] | 0.0 [0.0 to 7.9] | 2.3 [0.1 to 12.3] | 2.2 [0.1 to 11.5]
  Fever: >38.4 degrees C to 38.9 degrees C | 2.4 [0.1 to 12.9] | 0.0 [0.0 to 8.4] | 2.6 [0.1 to 13.5] | 0.0 [0.0 to 8.0] | 4.4 [0.5 to 15.1] | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 8.2] | 4.3 [0.5 to 14.8]
  Fever: >38.9 degrees C to 40.0 degrees C | 0.0 [0.0 to 8.6] | 2.4 [0.1 to 12.6] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 8.2] | 0.0 [0.0 to 7.7]
  Fever: >40.0 degrees C | 0.0 [0.0 to 8.6] | 0.0 [0.0 to 8.4] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 8.2] | 0.0 [0.0 to 7.7]
  Fatigue: Mild | 17.1 [7.2 to 32.1] | 19.0 [8.6 to 34.1] | 20.5 [9.3 to 36.5] | 13.6 [5.2 to 27.4] | 11.1 [3.7 to 24.1] | 21.7 [10.9 to 36.4] | 22.2 [11.2 to 37.1] | 20.9 [10.0 to 36.0] | 21.7 [10.9 to 36.4]
  Fatigue: Moderate | 14.6 [5.6 to 29.2] | 26.2 [13.9 to 42.0] | 12.8 [4.3 to 27.4] | 25.0 [13.2 to 40.3] | 31.1 [18.2 to 46.6] | 19.6 [9.4 to 33.9] | 11.1 [3.7 to 24.1] | 30.2 [17.2 to 46.1] | 15.2 [6.3 to 28.9]
  Fatigue: Severe | 0.0 [0.0 to 8.6] | 2.4 [0.1 to 12.6] | 0.0 [0.0 to 9.0] | 4.5 [0.6 to 15.5] | 4.4 [0.5 to 15.1] | 4.3 [0.5 to 14.8] | 2.2 [0.1 to 11.8] | 2.3 [0.1 to 12.3] | 8.7 [2.4 to 20.8]
  Headache: Mild | 34.1 [20.1 to 50.6] | 23.8 [12.1 to 39.5] | 25.6 [13.0 to 42.1] | 18.2 [8.2 to 32.7] | 13.3 [5.1 to 26.8] | 17.4 [7.8 to 31.4] | 15.6 [6.5 to 29.5] | 14.0 [5.3 to 27.9] | 13.0 [4.9 to 26.3]
  Headache: Moderate | 7.3 [1.5 to 19.9] | 11.9 [4.0 to 25.6] | 12.8 [4.3 to 27.4] | 9.1 [2.5 to 21.7] | 20.0 [9.6 to 34.6] | 6.5 [1.4 to 17.9] | 6.7 [1.4 to 18.3] | 14.0 [5.3 to 27.9] | 10.9 [3.6 to 23.6]
  Headache: Severe | 2.4 [0.1 to 12.9] | 0.0 [0.0 to 8.4] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 7.9] | 2.2 [0.1 to 11.5] | 0.0 [0.0 to 7.9] | 7.0 [1.5 to 19.1] | 0.0 [0.0 to 7.7]
  Muscle Pain: Mild | 12.2 [4.1 to 26.2] | 7.1 [1.5 to 19.5] | 12.8 [4.3 to 27.4] | 13.6 [5.2 to 27.4] | 8.9 [2.5 to 21.2] | 13.0 [4.9 to 26.3] | 2.2 [0.1 to 11.8] | 11.6 [3.9 to 25.1] | 17.4 [7.8 to 31.4]
  Muscle Pain: Moderate | 0.0 [0.0 to 8.6] | 14.3 [5.4 to 28.5] | 0.0 [0.0 to 9.0] | 9.1 [2.5 to 21.7] | 6.7 [1.4 to 18.3] | 13.0 [4.9 to 26.3] | 2.2 [0.1 to 11.8] | 18.6 [8.4 to 33.4] | 13.0 [4.9 to 26.3]
  Muscle Pain: Severe | 0.0 [0.0 to 8.6] | 2.4 [0.1 to 12.6] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.0] | 2.2 [0.1 to 11.8] | 4.3 [0.5 to 14.8] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 8.2] | 4.3 [0.5 to 14.8]
  Joint Pain: Mild | 2.4 [0.1 to 12.9] | 9.5 [2.7 to 22.6] | 5.1 [0.6 to 17.3] | 2.3 [0.1 to 12.0] | 6.7 [1.4 to 18.3] | 10.9 [3.6 to 23.6] | 4.4 [0.5 to 15.1] | 11.6 [3.9 to 25.1] | 2.2 [0.1 to 11.5]
  Joint Pain: Moderate | 0.0 [0.0 to 8.6] | 4.8 [0.6 to 16.2] | 0.0 [0.0 to 9.0] | 9.1 [2.5 to 21.7] | 4.4 [0.5 to 15.1] | 6.5 [1.4 to 17.9] | 0.0 [0.0 to 7.9] | 9.3 [2.6 to 22.1] | 13.0 [4.9 to 26.3]
  Joint Pain: Severe | 0.0 [0.0 to 8.6] | 0.0 [0.0 to 8.4] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 7.9] | 2.2 [0.1 to 11.5] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 8.2] | 2.2 [0.1 to 11.5]

3. Primary Outcome: Percentage of Participants With Adverse Events (AE) Within 1 Month After Administration of Study Intervention
Description: An AE was defined as any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. Exact 2-sided 95% CI was based on the Clopper and Pearson method.
Time Frame: Within 1 month after study intervention
Population: Safety population included all participants who received the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Candidate-1 | Candidate-2 | Candidate-3 | Candidate-4 | Candidate-5 | Candidate-6 | Candidate - Control | PCV15 | 13vPnC
Number analyzed (Participants) | 41 | 42 | 39 | 44 | 45 | 46 | 45 | 43 | 46
Percentage of participants | 2.4 [0.1 to 12.9] | 4.8 [0.6 to 16.2] | 5.1 [0.6 to 17.3] | 0.0 [0.0 to 8.0] | 8.9 [2.5 to 21.2] | 4.3 [0.5 to 14.8] | 0.0 [0.0 to 7.9] | 2.3 [0.1 to 12.3] | 2.2 [0.1 to 11.5]

4. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAE) Within 1 Month After Administration of Study Intervention
Description: An SAE was defined as any untoward medical occurrence that, at any dose, met one or more of the following criteria - resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect and was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic and other important medical event. Exact 2-sided 95% CI was based on the Clopper and Pearson method.
Time Frame: Within 1 month after study intervention
Population: Safety population included all participants who received the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Candidate-1 | Candidate-2 | Candidate-3 | Candidate-4 | Candidate-5 | Candidate-6 | Candidate - Control | PCV15 | 13vPnC
Number analyzed (Participants) | 41 | 42 | 39 | 44 | 45 | 46 | 45 | 43 | 46
Percentage of participants | 0.0 [0.0 to 8.6] | 0.0 [0.0 to 8.4] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 8.0] | 2.2 [0.1 to 11.8] | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 8.2] | 0.0 [0.0 to 7.7]

5. Secondary Outcome: Serotype Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) 1 Month After Administration of Study Intervention From Each Candidate and Candidate Control Group
Description: GMTs and the corresponding 2-sided CIs (from each candidate and candidate control group per the protocol objective) were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student's t distribution).
Time Frame: 1 month after study intervention
Population: Evaluable immunogenicity population included eligible participants who received study intervention as randomized, had at least 1 valid assay result within 27 to 49 days after administration, and had no major protocol deviations. Participants from each candidate and candidate control group were included as per the protocol specified objective. Number of Participants Analyzed= participants in evaluable immunogenicity population & had valid result 1 month after study intervention.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Candidate-1 | Candidate-2 | Candidate-3 | Candidate-4 | Candidate-5 | Candidate-6 | Candidate - Control
Number analyzed (Participants) | 41 | 42 | 38 | 43 | 43 | 45 | 43
Titer | 231 [162 to 328] | 428 [318 to 575] | 350 [254 to 481] | 354 [271 to 461] | 324 [239 to 439] | 536 [372 to 774] | 168 [116 to 244]

ADVERSE EVENTS:
Time Frame: Local reactions and systemic events (systematic assessment): up to 7 days after study intervention, SAEs (non-systemic assessment) and non-SAEs (systematic assessment): from Day 1 up to 1 month after study intervention.
Description: The same event may appear as both non-SAE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Safety population included all participants who received the study intervention.
Arm/Group | Candidate-1 | Candidate-2 | Candidate-3 | Candidate-4 | Candidate-5 | Candidate-6 | Candidate - Control | PCV15 | 13vPnC
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/42 | 0/39 | 0/44 | 0/45 | 0/46 | 0/45 | 0/43 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/42 | 0/39 | 0/44 | 1/45 | 0/46 | 0/45 | 0/43 | 0/46
Other Adverse Events (participants affected / at risk) | 25/41 | 27/42 | 21/39 | 28/44 | 30/45 | 30/46 | 22/45 | 32/43 | 37/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Candidate-1 (N=41) | Candidate-2 (N=42) | Candidate-3 (N=39) | Candidate-4 (N=44) | Candidate-5 (N=45) | Candidate-6 (N=46) | Candidate - Control (N=45) | PCV15 (N=43) | 13vPnC (N=46)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Candidate-1 (N=41) | Candidate-2 (N=42) | Candidate-3 (N=39) | Candidate-4 (N=44) | Candidate-5 (N=45) | Candidate-6 (N=46) | Candidate - Control (N=45) | PCV15 (N=43) | 13vPnC (N=46)
Fatigue (FATIGUE) (General disorders) | 13 | 20 | 13 | 19 | 21 | 21 | 16 | 23 | 21
Injection site erythema (REDNESS) (General disorders) | 0 | 1 | 0 | 1 | 2 | 3 | 0 | 4 | 1
Injection site pain (PAIN) (General disorders) | 5 | 13 | 8 | 12 | 20 | 19 | 6 | 29 | 29
Injection site swelling (SWELLING) (General disorders) | 0 | 1 | 1 | 1 | 2 | 4 | 0 | 4 | 4
Pyrexia (FEVER) (General disorders) | 1 | 1 | 1 | 0 | 3 | 2 | 0 | 1 | 3
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 1 | 6 | 2 | 5 | 5 | 9 | 2 | 9 | 8
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 5 | 10 | 5 | 10 | 8 | 14 | 2 | 13 | 16
Headache (HEADACHE) (Nervous system disorders) | 18 | 15 | 15 | 12 | 15 | 12 | 10 | 15 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT05489328/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/28/NCT05489328/SAP_001.pdf